CLINICAL TRIAL: NCT04008966
Title: Comparative Study Between Single Versus Dual Trigger for Poor Responders in GnRH-antagonist ICSI Cycles. A Randomized Controlled Study
Brief Title: Comparative Study Between Single Versus Dual Trigger for Poor Responders in GnRH-antagonist ICSI Cycles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 58
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Assisted Reproduction
MeSH Terms: interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; cetrorelix; Chorionic Gonadotropin; Gonadotropin-Releasing Hormone; Triptorelin Pamoate; Embryo Transfer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single trigger (Active Comparator): 80 women who received triggering in the form of 10,000 IU of HCG intramuscular injection
  Interventions: Drug: combined oral contaraceptive pills; Drug: recombinant FSH; Drug: Urinaru gonadotropin; Drug: GnRH antagonist; Drug: Human chorionic gonadotropin; Procedure: Ovum pick up; Procedure: Embryo transfer; Drug: natural Progesterone
- Dual trigger (Active Comparator): 80 women who received triggering in the form of 10,000 IU of HCG intramuscular injection in addition to GnRH agonist triptorelin 0.2 mg subcutaneously
  Interventions: Drug: combined oral contaraceptive pills; Drug: recombinant FSH; Drug: Urinaru gonadotropin; Drug: GnRH antagonist; Drug: Human chorionic gonadotropin; Drug: GnRH agonist; Procedure: Ovum pick up; Procedure: Embryo transfer; Drug: natural Progesterone

INTERVENTIONS:
Drug: combined oral contaraceptive pills — 1 tablet daily between days 5 and 25 of the cycle before stimulation
  Other Names: Gynera
Drug: recombinant FSH — 300 U from the 2nd day of the cycle then the dose was adjusted according to the ovarian response evaluated by transvaginal ultrasound and serum E2
Drug: Urinaru gonadotropin — 150 U from the 2nd day of the cycle then the dose was adjusted according to the ovarian response evaluated by transvaginal ultrasound and serum E2
Drug: GnRH antagonist — 0.25 subcutaneously daily from the day in which the leading follicles reached 12 mm till the day of triggering
  Other Names: Cetrotide
Drug: Human chorionic gonadotropin — 10,000 IU intramuscular when at least 3 follicles larger than 14 mm and at least one of them reached a mean diameter of 17 mm or more
Drug: GnRH agonist — 0.2 mg subcutaneously when at least 3 follicles larger than 14 mm and at least one of them reached a mean diameter of 17 mm or more
  Other Names: triptorelin
  Arms: Dual trigger
Procedure: Ovum pick up — 34 hours after triggering under the guidance of transvaginal ultrasound
Procedure: Embryo transfer — Transabdominal ultrasound guided embryo transfer was done 3 days after oocyte retrieval using Labotect semirigid catheter
Drug: natural Progesterone — 400 mg twice daily per vagina
  Other Names: Prontogest

SUMMARY:
All participants started with a combination of recombinant FSH 300 U and urinary Gn 150 U from the 2nd day of the cycle then the dose was adjusted according to the ovarian response

From day 6 of the cycle, follow up using transvaginal ultrasound was done either daily or on alternate days according to the ovarian response. When the leading follicle reached 12 mm, GnRH antagonist was started using Cetrotide 0.25 subcutaneously daily till the day of triggering. Triggering was done when at least 3 follicles larger than 14 mm and at least one of them reached a mean diameter of 17 mm or more.

At the day of triggering, women were randomized into 2 groups. Group I (single trigger group) that included 80 women who received triggering in the form of 10,000 IU of HCG intramuscular injection. Group II (Dual trigger group) that included 80 women who received triggering in the form of 10,000 IU of HCG intramuscular injection in addition to GnRH agonist triptorelin 0.2 mg subcutaneously.

Ovum pickup was done 34 hours after triggering under the guidance of transvaginal ultrasound.

ISM1 culture medium was used for oocyte collection and embryo culture. Transabdominal ultrasound guided embryo transfer was done 3 days after oocyte retrieval using Labotect semirigid catheter by the same expert operator

Cycle cancellation was done if day 9 folliculometry revealed less than 2 mature follicles, no oocytes were retrieved or if fertilization failed

Luteal phase support was started in all women on the day of oocyte retrieval and continued till the day of serum β-hCG assessment (done 14 days after ET) through administration of 400 mg of natural Progesterone twice daily per vagina . In women with +ve serum β-hCG (> 5 mIU/ml), transvaginal ultrasound evaluation was done 4 weeks after ET to confirm the presence and number of intrauterine gestational sacs.

DETAILED DESCRIPTION:
All participants started with a combination of recombinant FSH 300 U and urinary Gn 150 U from the 2nd day of the cycle then the dose was adjusted according to the ovarian response evaluated by transvaginal ultrasound and serum E2. Delayed start

From day 6 of the cycle, follow up using transvaginal ultrasound was done either daily or on alternate days according to the ovarian response. Ultrasound follow up reported number and size of follicles in each ovary and the endometrial thickness and pattern. When the leading follicle reached 12 mm, GnRH antagonist was started using Cetrotide 0.25 subcutaneously daily till the day of triggering. Triggering was done when at least 3 follicles larger than 14 mm and at least one of them reached a mean diameter of 17 mm or more.

At the day of triggering, women were randomized into 2 groups. Group I (single trigger group) that included 80 women who received triggering in the form of 10,000 IU of HCG intramuscular injection. Group II (Dual trigger group) that included 80 women who received triggering in the form of 10,000 IU of HCG intramuscular injection in addition to GnRH agonist triptorelin 0.2 mg subcutaneously.

Ovum pickup was done 34 hours after triggering under the guidance of transvaginal ultrasound.

ISM1 culture medium was used for oocyte collection and embryo culture. Transabdominal ultrasound guided embryo transfer was done 3 days after oocyte retrieval using Labotect semirigid catheter by the same expert operator

Cycle cancellation was done if day 9 folliculometry revealed less than 2 mature follicles, no oocytes were retrieved or if fertilization failed

Luteal phase support was started in all women on the day of oocyte retrieval and continued till the day of serum β-hCG assessment (done 14 days after ET) through administration of 400 mg of natural Progesterone twice daily per vagina . In women with +ve serum β-hCG (> 5 mIU/ml), transvaginal ultrasound evaluation was done 4 weeks after ET to confirm the presence and number of intrauterine gestational sacs.

ELIGIBILITY:
Inclusion Criteria:

* women with poor ovarian response candidate for ICSI
* women with spontaneous normal menstrual cycle
* normal uterine cavity

Exclusion Criteria:

* women with ovarian cysts
* endometriosis
* hydrosalpinx
* endocrinological disorders as hyperprolactinemia, thyroid or adrenal disorders.
* Couples with azospermic male partner
* those with severe uncontrolled medical or metabolic disorders

Ages: 25 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 160 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2019-06-02 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
number of mature follicular count | 10 - 14 days of the cycle
  number of follicles larger than 14 mm

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed maged, MD, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

REFERENCES:
- [Derived] Maged AM, Ragab MA, Shohayeb A, Saber W, Ekladious S, Hussein EA, El-Mazny A, Hany A. Comparative study between single versus dual trigger for poor responders in GnRH-antagonist ICSI cycles: A randomized controlled study. Int J Gynaecol Obstet. 2021 Mar;152(3):395-400. doi: 10.1002/ijgo.13405. Epub 2020 Oct 22. PMID 33011968